CLINICAL TRIAL: NCT00575887
Title: Efficacy of a Protracted Temozolomide Schedule in Patients With Progression After Standard Dose Temozolomide for High-grade Gliomas
Brief Title: Efficacy of Protracted Temozolomide in Patients With Progressive High Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Principal Investigator, Ufuk ABACIOGLU, Assoc. Prof., Marmara University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MU-RO-2005-1
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-11

CONDITIONS: Glioblastoma; Astrocytoma; Oligodendroglioma; Brain Tumor, Recurrent
Keywords: Temozolomide; Brain Tumor, Recurrent; Chemotherapy
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — 100 mg/m2/day, (PO) orally, on days between 1 and 21 of each 28 day cycles. Number of cycles: Until progression or unacceptable toxicity
  Other Names: Temodal; Temodar

SUMMARY:
The purpose of this study is to evaluate the efficacy of temozolomide on a protracted schedule, after standard 5-day temozolomide regimen in patients with recurrent or progressive high grade glioma.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18 years old
* Histopathological diagnosis of high grade glioma (anaplastic astrocytoma or anaplastic oligodendroglioma or anaplastic oligoastrocytoma or glioblastoma multiforme)
* Progression after standard dose (D1-5/28 days)temozolomide either during recurrence or adjuvant treatment approved in Magnetic Resonance imaging
* Karnofsky Performance Status scale >/=50 (due to brain pathology)
* Adequate hematological, renal and hepatic function
* Patients willing to participate in the study and signing the informed consent

Exclusion Criteria:

* Karnofsky Performance Status scale <50
* Female patients with pregnancy or with suspicion of pregnancy. Patients with fertility will be warned for appropriate contraception during the study
* Patients not suitable for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk ABACIOGLU, MD, Study Chair — Marmara University Hospital, Radiation Oncology Department
Locations (1):
- Marmara University Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Abacioglu U, Caglar HB, Yumuk PF, Akgun Z, Atasoy BM, Sengoz M. Efficacy of protracted dose-dense temozolomide in patients with recurrent high-grade glioma. J Neurooncol. 2011 Jul;103(3):585-93. doi: 10.1007/s11060-010-0423-2. Epub 2010 Sep 29. PMID 20878446

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose-Dense Temozolomide: Temozolomide : 100 mg/m2/day, (PO) orally, on days between 1 and 21 of each 28 day cycles.
  Number of cycles: Until progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Dose-Dense Temozolomide
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dose-Dense Temozolomide
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 50 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Region of Enrollment [Number; unit: participants]
  Turkey | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6-months
Time Frame: Until progression
Measure: Number; unit: percentage of participants
Groups:
- Temozolomide: Temozolomide : 100 mg/m2/day, (PO) orally, on days between 1 and 21 of each 28 day cycles.
  Number of cycles: Until progression or unacceptable toxicity
Arm/Group | Temozolomide
Number analyzed (Participants) | 25
percentage of participants | 17.3

ADVERSE EVENTS:
Arm/Group | Temozolomide
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 20/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=25)
Lymphopenia (Blood and lymphatic system disorders) | 20 (20) — Gr 3-4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) — Gr 3-4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No